CLINICAL TRIAL: NCT02615275
Title: Validation of Eight-Electrode Multifrequency Bioelectrical Impedance Analysis to Estimate Body Composition in a Head and Neck Cancer Population Undergoing Radiation Therapy
Brief Title: Bioelectrical Impedance Analysis in Estimating Body Composition in Patients With Stage I-IV Head and Neck Cancer Undergoing Radiation Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA15-0600; NCI-2018-02603 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA15-0600 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Carcinoma
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (bioelectrical impedance analysis, RT) (Experimental): Patients undergo bioelectrical impedance analysis with seca mBCA and CT or PET at baseline, weekly for 6-7 weeks during standard of care RT, and at 10-12 weeks after completion of RT.
  Interventions: Procedure: Bioelectric Impedance Analysis; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Bioelectric Impedance Analysis — Undergo BIA with seca mBCA
  Other Names: BIA; Bioelectric Impedance; Bioelectric Impedance Test; Bioelectrical Impedance Analysis; Bioimpedance Analysis
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation

SUMMARY:
Bioelectrical impedance analysis measures body mass (the amount of muscle and fat in the body) and the level of hydration to help researchers identify patients who are losing muscle mass during radiation therapy. This information may help researchers make decisions about nutritional supplementation and the placement of feeding tubes in patients receiving radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To validate body composition estimates derived from the seca (SECA) medical body composition analyzer (mBCA) bioelectrical impedance analysis (BIA) scale by comparing with computed tomography (CT) measured lean and fat body mass.

SECONDARY OBJECTIVES:

I. Evaluate sensitivity of mBCA to detect changes in body composition during treatment.

II. Identify whether BIA-estimated loss of lean body mass (LBM) during treatment predicts development of sarcopenia.

III. Determine whether BIA-derived estimates of body water correlate with requirements for intravenous (IV) hydration and unplanned hospital admissions.

IV. Explore associations between body composition and symptom burden during treatment.

OUTLINE:

Patients undergo bioelectrical impedance analysis with seca mBCA and CT or positron emission tomography (PET) at baseline, weekly for 6-7 weeks during standard of care radiation therapy (RT), and at 10-12 weeks after completion of RT.

After completion of study, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented head and neck cancer (clinical stage I-IVB; Tx,1-4, N0-3).
* Patients dispositioned to receive radiation therapy (dose >= 60 gray [Gy]).
* Patients may receive radiation as either primary therapy or post-operatively.
* Patient received staging positron emission tomography/computed tomography (PET/CT) scan during 60-day period prior to initiating therapy.
* Negative pregnancy test for women of child bearing potential.

Exclusion Criteria:

* Previous radiation treatment for head and neck mucosal primary cancers (i.e. oropharynx, nasopharynx, hypopharynx, larynx, and oral cavity).
* Patients with pacemaker, implanted cardiac defibrillator, or vagal nerve stimulator.
* Pregnant or breast-feeding females.
* Patients weighing over 660 lbs (300 kg).
* Patients with other medical conditions known to cause sarcopenia, including New York Heart Association (NYHA) class III-IV heart failure, oxygen-dependent pulmonary disease, advanced human immunodeficiency virus infection, cirrhosis, end stage renal disease, or inherited/congenital disorders of metabolism.
* Patients receiving palliative irradiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Lean and Fat Body Mass Composition from SECA mBCA BIA Scale Compared with Computed Tomography (CT) in Participants with Head and Neck Cancer Undergoing Radiation Therapy (RT) | 7 weeks
  Validation of BIA measures of body composition made by comparison with CT-based estimates of body composition.
  Linear regression analysis used to determine the relative agreement between lean body mass and fat body mass predicted from impedance measurement and CT imaging.

SECONDARY OUTCOMES:
BIA-derived body composition calculations | Up to 2 years
  Root mean square error analysis will be utilized to quantify the average error from BIA-derived body composition calculations.

OTHER OUTCOMES:
Bioelectrical impedance analysis (BIA) estimates of total body water | Up to 2 years
  a. Bioelectrical impedance analysis (BIA) estimates of total body water (kg)
The incidence of unplanned hospitalizations | Up to 2 years
  b. incidence of unplanned hospitalizations (#)
Lean body mass as a predictor of sarcopenia | Up to 2 years
  Exploratory analyses will evaluate whether decreases in lean mass measured during treatment correlates to the presence of sarcopenia on follow up.
Lean body mass as a predictor of therapeutic feeding tube use | Up to 2 years
  Exploratory analyses will evaluate whether decreases in lean mass measured during treatment correlates to the incidence of therapeutic feeding tube use.
Quality of life assessed questionnaire | Baseline up to 12 months
  a. MD Anderson Symptom Inventory-Head and Neck (MDASI-HN)
Quality of life questionnaire | Baseline up to 12 months
  b. Brief patient interviews to assess performance status (ECOG PS) Scores 0-5

CONTACTS AND LOCATIONS:
Overall Officials: Clifton D Fuller, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org